CLINICAL TRIAL: NCT02892227
Title: Management of Acute Heart Failure: Contribution of Ultrasound Daily "in Bed Patient" Adjustment on Therapy With Impact Measure on re Hospital Rate During 30 Days
Acronym: JECICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOI/2015/JER-01; 2016-A00635-46 (Other: ANSM)
Record Dates: First submitted 2016-08-26; First posted 2016-09-08 (Estimated); Last update posted 2025-12-01 (Actual); Status verified 2018-12

CONDITIONS: Heart Failure
Keywords: bedside echography
MeSH Terms: conditions — Heart Failure

ARMS (2):
- JET ECHO (Experimental): Transmitral flow estimation
  Interventions: Procedure: Transmitral flow estimation
- NO JET ECHO (No Intervention): no bedside echocardiography

INTERVENTIONS:
Procedure: Transmitral flow estimation — Estimation of the transmitral flow of the inferior vena cava and its variations
  Arms: JET ECHO

SUMMARY:
Our hypothesis: a daily bedside echocardiographic assessment, protocolized, simple and reproducible estimation of filling pressures with an evaluation of mitral inflow and the inferior vena cava, allow a more reliable estimate of the true blood volume of the patient and thus lead to a therapeutic adjustment more suitable.

This therapeutic adjustment closer to patient's needs would impact fewer readmissions at 30 days and mortality, less alteration of biological parameters myocardial, kidney and liver.

ELIGIBILITY:
Inclusion Criteria:

The patient or his representative must be given free and informed consent and signed consent.

* The patient must be affiliated or beneficiary of a health insurance plan.
* The patient is available for a follow-up 6 months.
* The patient is of age or older (>) 18.
* Patients hospitalized for acute heart failure who received at least 40mg of furosemide IV.
* Patient with impaired LVEF <50%.
* Patient with Nt-proBNP values> 1200pg / ml.

Exclusion Criteria:

* The subject takes part in another study.

  * The subject is exclusion period determined by a previous study.
  * The subject is under judicial protection.
  * The subject or his representative refuses to sign the consent.
  * It is not possible to give the subject or his representative informed information.

Non-inclusion criteria for those diseases or conditions associated (s) interfere (s):

* The patient is pregnant or is breastfeeding.
* The patient is already included in a surveillance program (PRADO, OSICAT).
* Patient with a mechanical or biological mitral prosthesis.
* History of mitral stenosis.
* severe valvular surgery with maturity in months (<30 days).
* chronic renal impairment on dialysis.
* High grade AV block (AVB and BAV3 2/1).
* Hypertrophic cardiomyopathy.
* Cardiogenic shock.
* Contraindications to furosemide.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
rehospitalization | 30 days

SECONDARY OUTCOMES:
mortality | 6 months
worsening heart failure | during hospitalization
average length of stay | during hospitalization
alteration of biological parameters myocardial, kidney and liver | Hospital discharge +7 days, Hospital discharge +30 days

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Arnaud de Villeneuve, Montpellier
  - CHU Nimes, Nîmes

REFERENCES:
- [Result] Ricci JE, Aguilhon S, Occean BV, Soullier C, Solecki K, Robert C, Huet F, Cornillet L, Schmutz L, Chevallier T, Akodad M, Leclercq F, Cayla G, Lattuca B, Roubille F. Impact of Daily Bedside Echocardiographic Assessment on Readmissions in Acute Heart Failure: A Randomized Clinical Trial. J Clin Med. 2022 Apr 6;11(7):2047. doi: 10.3390/jcm11072047. PMID 35407655